CLINICAL TRIAL: NCT04202549
Title: Improving Neuroprotective Strategy for Ischemic Stroke With Sufficient Recanalization After Thrombectomy by Intra-arterial Cocktail Therapy (INSIST-CT): a Prospective, Single Arm, Pilot Study
Brief Title: Improving Neuroprotective Strategy for Ischemic Stroke With Sufficient Recanalization After Thrombectomy by Intra-arterial Cocktail Therapy (INSIST-CT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hui-Sheng Chen (Other)
Responsible Party: Sponsor-Investigator, Hui-Sheng Chen, Professor, General Hospital of Shenyang Military Region
Organization: General Hospital of Shenyang Military Region (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: k(2019)31
Record Dates: First submitted 2019-12-15; First posted 2019-12-17 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intra-arterial cocktail therapy (Experimental): Intra-arterial administration of argatroban (0.2-0.3 mg/min), dexamethasone (0.1 mg/min) and edaravone (0.3 mg/min) for 30 to 60 minutes after thrombectomy
  Interventions: Drug: intra-arterial cocktail therapy

INTERVENTIONS:
Drug: intra-arterial cocktail therapy — Intra-arterial administration of argatroban (0.2-0.3 mg/min), dexamethasone (0.1 mg/min) and edaravone (0.3 mg/min) for 30 to 60 minutes after thrombectomy.

SUMMARY:
Thrombolysis and endovascular thrombectomy are the most efficient treatments for acute ischemic stroke patients in time window. Although sufficient recanalization after thrombectomy is more than 80%, HERMES study indicated that nearly half of the ischemic stroke patients under thrombectomy suffered obvious disability. Artery reocclusion, hemorrhagic transformation, and no-reflow phenomenon are among the most important reasons of poor prognosis of acute ischemic stroke patients. The investigators speculate that a combination of argatroban, edaravone, and glucocorticoid may be helpful in preventing artery reocclusion, hemorrhagic transformation, and no-reflow phenomenon. This study intends to explore the safety, feasibility and efficacy of thrombectomy with sufficient recanalization bridged by intra-arterial cocktail therapy in acute ischemic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Patients who presented with acute ischemic stroke and a large vessel occlusion in the anterior circulation and met the criteria of mechanical thrombectomy.
3. Sufficient recanalization （TICI 2b-3）within 7 hours of stroke onset.
4. The availability of informed consent.

Exclusion Criteria:

1. insufficient recanalization（TICI < 2a）after endovascular treatment;
2. Hemorrhagic stroke: cerebral hemorrhage, subarachnoid hemorrhage.

4. Coagulation disorders, systematic hemorrhagic tendency, thrombocytopenia （ <100000/mm3）.

5. Severe hepatic or renal dysfunction, increase in ALT or AST (more than 2 times of upper limit of normal value), increase in serum creatinine (more than 1.5 times of upper limit of normal value) or requiring dialysis.

6. Severe uncontrolled hypertension (systolic blood pressure over 200mmHg or diastolic blood pressure over 110 mmHg).

7. Patients with contraindication or allergic to any ingredient of drugs in our study.

8. Unsuitable for this clinical studies assessed by researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Proportion of favorable outcome | 90 days
  favorable outcome is defined as mRS 0-2

SECONDARY OUTCOMES:
Proportion of excellent outcome | 90 days
  excellent outcome is defined as mRS 0-1
proportion of early neurological improvement | 48 hours
  early neurological improvement is defined as more than 4 decrease in NIHSS

OTHER OUTCOMES:
incidence of symptomatic intracranial haemorrhage | 48 hours
  intracranial haemorrhage is defined as more than 4 increase in NIHSS caused by intracranial bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, China

REFERENCES:
- [Derived] Zhao ZA, Hu HZ, Li W, Qiu J, Zhao YG, Nguyen TN, Chen HS. Intra-arterial cocktail therapy for patients with anterior circulation large vessel occlusion who achieved endovascular reperfusion. Front Neurol. 2024 Dec 6;15:1450156. doi: 10.3389/fneur.2024.1450156. eCollection 2024. PMID 39711792